CLINICAL TRIAL: NCT06746896
Title: A Retrospective Study on the Role of Short-chain Fatty Acids Modulation in Multiple Sclerosis
Brief Title: Retrospective Study on the Role of SCFA Modulation in Multiple Sclerosis
Status: Active, not recruiting | Type: Observational
Sponsor: Prof. Massimo Filippi (Other)
Collaborators: Università Vita-Salute San Raffaele (Other)
Responsible Party: Sponsor-Investigator, Prof. Massimo Filippi, Prof., IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: Brainess FISM
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Gut-brain axis; SCFA; Microbiota
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Urines, plasma, CSF, stool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Controls: Absence of neurological symptoms or known diagnosis, absence of a known gastrointestinal pathology.
- Newly diagnosed MS patients: Absence of a known gastrointestinal pathology.

SUMMARY:
Recent studies show that gut microbiota strongly influences multiple sclerosis. These data suggest that the microbiota could have a direct effect on MS pathogenesis, although the mechanisms through which it modulates central nervous system (CNS) neuroinflammation and neurodegeneration are still poorly defined. The microbiota mediates its action principally through synthesizing specific metabolites that act as messengers in host functions, such as the modulation of the immune and nervous system, tissue repair, and stemness. The short-chain fatty acids (SCFAs- mainly acetate, propionate, and butyrate), produced by the fermentation of dietary fibers, are a class of microbial metabolites of primary importance for host physiology. Thus, the objective is to establish a mechanistic link between gut microbiota dysbiosis, reflected by a different level of SCFAs and SCFA-producing bacteria species, and neuroimmune alterations in MS. Preliminary data show a differential metabolomic profile in urine samples of MS patients compared to healthy controls. The authors now aim at deepening previous findings by analysing also the SCFAs concentration in the urines, plasma and CSF by GC-MS (their level turned out to be too low to be measured by NMR) and the microbiota composition by shotgun metagenomics analysis, to track changes in the abundance of SCFAs-producing bacteria species.

ELIGIBILITY:
Inclusion Criteria:

- Volunteers that have preventively signed the informed consent to use their samples for additional studies.

Exclusion Criteria:

- None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 healthy controls and 20 newly diagnosed not yet treated MS patients. Both HC and MS were recruited inside IRCCS San Raffaele. Both categories are composed of 50% females and 50% males. The age range for both categories is comprised between 28 and 65 years.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Modulation of SCFAs levels in MS patients versus healthy controls. | Baseline
  Quantification of SCFAs (mainly acetate, butyrate and propionate) in different biofluids and samples: urines, plasma and CSF. It will be obtained by GC-MS.

SECONDARY OUTCOMES:
Gut microbial composition in MS patients versus healthy controls | Baseline
  To perform taxonomical and functional analysis of the intestinal microbiota. We will examine bacteria DNA from stool samples by shotgun metagenomic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy, Italy

REFERENCES:
- [Background] Duscha A, Gisevius B, Hirschberg S, Yissachar N, Stangl GI, Dawin E, Bader V, Haase S, Kaisler J, David C, Schneider R, Troisi R, Zent D, Hegelmaier T, Dokalis N, Gerstein S, Del Mare-Roumani S, Amidror S, Staszewski O, Poschmann G, Stuhler K, Hirche F, Balogh A, Kempa S, Trager P, Zaiss MM, Holm JB, Massa MG, Nielsen HB, Faissner A, Lukas C, Gatermann SG, Scholz M, Przuntek H, Prinz M, Forslund SK, Winklhofer KF, Muller DN, Linker RA, Gold R, Haghikia A. Propionic Acid Shapes the Multiple Sclerosis Disease Course by an Immunomodulatory Mechanism. Cell. 2020 Mar 19;180(6):1067-1080.e16. doi: 10.1016/j.cell.2020.02.035. Epub 2020 Mar 10. PMID 32160527